CLINICAL TRIAL: NCT06564454
Title: Assessment of Knowledge, Attitude and Practices Regarding Green Eco-Friendly Dentistry Among a Group of Dentists: A Cross-Sectional Study
Brief Title: Knowledge, Attitude and Practices Regarding Green Eco-Friendly Dentistry Among a Group of Dentists
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Abdelgawad, Associate Professor, Cairo University
Other Study IDs: CEBD-CU-2024-08-15
Record Dates: First submitted 2024-08-15; First posted 2024-08-21 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: Green Dentistry; Eco-friendly Dentistry; Knowledge; Attitude; Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: No intervention — Assessment of knowledge, attitude and practice of green Dentistry

SUMMARY:
Global warming, reduction in resources, increase in prices are all factors leading to more direction towards reuse, recycling, and reduction in use of materials. The World Dental Federation (FDI) considers sustainability to be an indispensable principle of Dentistry, which "must be practiced ethically, with high levels of quality and safety, in the pursuit of optimal oral health. Sustainability requires more attention from dental health professionals to reduce, recycle and reuse available resources.

DETAILED DESCRIPTION:
The direction towards more reuse, recycling and reduction in the use of materials is a global direction. The Egyptian society needs to address the concepts, however, there is lack of knowledge on the knowledge, attitude, and practices of Egyptian dentists regarding green eco-friendly Dentistry.

Research question:

What is the knowledge, attitude, and practices of a group of dentists regarding green eco-friendly Dentistry?

ELIGIBILITY:
Inclusion Criteria:

* Graduated dentists.
* Dentists graduated from Egyptian universities.

Exclusion Criteria:

* Refusal of participation.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Graduated dentists.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Knowledge, attitude, and practices regarding green eco-friendly Dentistry. | Immediately after the dentists complete the questionnaire
  Knowledge, attitude, and practices of dentists regarding green eco-friendly Dentistry using a validated questionnaire, the unit is percentage of participants answering each question.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided